CLINICAL TRIAL: NCT04016805
Title: A Phase 2 Study to Assess the Efficacy and Safety of Ublituximab and Umbralisib in Subjects With Chronic Lymphocytic Leukemia (CLL) Currently Treated With Ibrutinib, Acalabrutinib or Venetoclax
Brief Title: Study to Assess the Efficacy and Safety of Ublituximab and Umbralisib in Participants With Chronic Lymphocytic Leukemia (CLL) Currently Treated With Ibrutinib, Acalabrutinib or Venetoclax
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic/Business decision
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTX-TGR-208
Record Dates: First submitted 2019-07-10; First posted 2019-07-11 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: umbralisib; ublituximab; venetoclax; ibrutinib; CLL; acalabrutinib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ublituximab; umbralisib; ibrutinib; venetoclax; acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ublituximab + umbralisib + ibrutinib (Experimental): Participants were administered with ublituximab, 900 milligrams (mg), intravenous (IV) infusion once every cycle through cycle 6, then every three cycles upto 24 cycles; umbralisib, 800 mg, oral tablet, daily through Cycles 1-24; ibrutinib oral tablet daily (1 Cycle = 28 days).
  Interventions: Drug: Ublituximab; Drug: Umbralisib; Drug: Ibrutinib
- ublituximab + umbralisib + venetoclax (Experimental): Participants were administered with ublituximab, 900 milligrams (mg), intravenous (IV) infusion once every cycle through cycle 6, then every three cycles upto 24 cycles; umbralisib, 800 mg, oral tablet, daily through Cycles 1-24; venetoclax oral tablet daily (1 Cycle = 28 days).
  Interventions: Drug: Ublituximab; Drug: Umbralisib; Drug: Venetoclax
- ublituximab + umbralisib + acalabrutinib (Experimental): Participants were administered with ublituximab, 900 milligrams (mg), intravenous (IV) infusion once every cycle through cycle 6, then every three cycles upto 24 cycles; umbralisib, 800 mg, oral tablet, daily through Cycles 1-24; acalabrutinib oral capsule every 12 hours (1 Cycle = 28 days).
  Interventions: Drug: Ublituximab; Drug: Umbralisib; Drug: Acalabrutinib Oral Capsule

INTERVENTIONS:
Drug: Ublituximab — * recombinant chimeric anti-CD20 monoclonal antibody
  * administered as an IV infusion
  Other Names: TG-1101
Drug: Umbralisib — * Phosphoinositide-3-kinase (PI3K) delta inhibitor
  * Tablet form, to taken orally on a daily basis
  Other Names: TGR-1202
Drug: Ibrutinib — * Bruton Tyrosine Kinase (BTK) inhibitor
  * Tablet form, to taken orally on a daily basis
  Other Names: Imbruvica
  Arms: ublituximab + umbralisib + ibrutinib
Drug: Venetoclax — * BCL-2 inhibitor
  * Tablet form, to be taken orally
  Other Names: Venclexta
  Arms: ublituximab + umbralisib + venetoclax
Drug: Acalabrutinib Oral Capsule — Kinase inhibitor, capsule form, to be taken orally
  Other Names: Calquence
  Arms: ublituximab + umbralisib + acalabrutinib

SUMMARY:
Phase 2, two cohort trial evaluating the addition of ublituximab and umbralisib on the rate of minimal residual disease (MRD) negativity in participants with Chronic Lymphocytic Leukemia (CLL), who are currently on treatment with ibrutinib, alacabrutinib or venetoclax.

DETAILED DESCRIPTION:
This is a Phase 2 open label, two treatment cohort trial evaluating the addition of ublituximab and umbralisib on the rate of minimal residual disease (MRD) negativity in participants with CLL, who fail to achieve MRD negativity, after a minimum 6-month treatment with ibrutinib, alacabrutinib or venetoclax.

ELIGIBILITY:
Inclusion Criteria:

* Participants with Chronic Lymphocytic Leukemia (CLL) who have been on treatment for at least 6 months
* Minimal Residual Disease positive at screening
* Adequate organ system function as specified in the protocol
* Ability to follow protocol procedures.

Exclusion Criteria:

* Participants receiving cancer therapy or any investigational drug within 21 days of Cycle 1, Day 1.
* Participants with a known histological transformation
* Active Hepatitis B or Hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2022-05-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - TG Therapeutics Investigational Trial Site, Boston, Massachusetts
  - TG Therapeutics Investigational Trial Site, Hackensack, New Jersey
  - TG Therapeutics Investigational Trial Site, New York, New York

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 41 participants were enrolled at 8 investigative sites across United States.
Period: Overall Study
Arm/Group | Ublituximab + Umbralisib + Ibrutinib | Ublituximab + Umbralisib + Venetoclax | Ublituximab + Umbralisib + Acalabrutinib
Started | 30 | 6 | 5
Completed | 0 | 0 | 0
Not Completed | 30 | 6 | 5
Not completed — Sponsor's Discretion | 30 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ublituximab + Umbralisib + Ibrutinib | Ublituximab + Umbralisib + Venetoclax | Ublituximab + Umbralisib + Acalabrutinib | Total
Number analyzed (Participants) | 30 | 6 | 5 | 41
Age, Continuous [Median (Full Range); unit: years] | 63 [48 to 81] | 54.5 [41 to 67] | 71 [57 to 77] | 63 [41 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 0 | 8
  Male | 23 | 5 | 5 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Rate of Undetected Minimal Residual Disease (U-MRD)
Description: U-MRD rate was defined as the proportion of participants who have undetectable MRD in the peripheral blood as confirmed by central lab.
Time Frame: Up to approximately 23 months
Population: Data for this outcome measure was not collected or analyzed as planned as the study was terminated due to sponsor's business decision.
Arm/Group | Ublituximab + Umbralisib + Ibrutinib | Ublituximab + Umbralisib + Venetoclax | Ublituximab + Umbralisib + Acalabrutinib
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as percent of participants who achieve complete response (CR) or partial response (PR). CR was defined as no evidence of new disease, regression of all target nodal masses to normal size < or = 1.5 cm in the longest diameter (LD) and an absolute lymphocyte count (ALC) in peripheral blood < 4*10^9/L. PR was defined as no evidence of new disease, a decrease in peripheral blood ALC by ≥50% from baseline or a decrease to <4 x 10^9/L or a decrease by ≥50% from the baseline in the sum of the products (SPD) of the target nodal lesions or a decrease by ≥50% from baseline in the CLL marrow infiltrate or in B lymphoid, no target, splenic, liver, or non-target disease with worsening that meets the criteria for definitive nodules, peripheral blood counts with ANC >1.5 x 10^9/L or platelet count ≥100 x 10^9/L or hemoglobin ≥110 g/L (11.0 g/dL) without red blood cell transfusions, all without need for exogenous growth factors.
Time Frame: Up to approximately 34 months
Population: as for outcome 1
Arm/Group | Ublituximab + Umbralisib + Ibrutinib | Ublituximab + Umbralisib + Venetoclax | Ublituximab + Umbralisib + Acalabrutinib
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) as Assessed by National Cancer Institute - Common Terminology Criteria for Adverse Events-Version (NCI-CTCAE-V5)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product. An AE does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. A TEAE is an AE that starts or worsens after receiving study drug.
Time Frame: Up to approximately 34 months
Population: as for outcome 1
Arm/Group | Ublituximab + Umbralisib + Ibrutinib | Ublituximab + Umbralisib + Venetoclax | Ublituximab + Umbralisib + Acalabrutinib
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: No safety data was collected and analyzed as planned at the end of study
Description: Study was terminated due to sponsor's business decision. Hence, no safety data was collected and analyzed as planned at the end of study
Arm/Group | Ublituximab + Umbralisib + Ibrutinib | Ublituximab + Umbralisib + Venetoclax | Ublituximab + Umbralisib + Acalabrutinib
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Due to sponsor's business decision, the clinical trial was terminated by the sponsor prematurely. No analysis was done at the termination of the trial, therefore, outcome, and safety data are not available and the numbers of participants analyzed are reported as "0".

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT04016805/Prot_SAP_000.pdf